CLINICAL TRIAL: NCT03126994
Title: Prospective, Single-Center, Non-Randomized Study of the PhysioWave™ Cardiovascular Analyzer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PhysioWave, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 780-00033
Record Dates: First submitted 2017-04-10; First posted 2017-04-25 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Cardiovascular Risk Factor
MeSH Terms: interventions — Pulse Wave Analysis

STUDY DESIGN:
Intervention Model Description: Prospective validation study to evaluate PWV, PR, and BW accuracy in a sample of subjects representing the US general adult population.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- PhysioWave Cardiovascular Analyzer (Experimental): The Experimental Device is the PhysioWave Cardiovascular Analyzer, which will be used to measure Pulse Wave Velocity, Pulse Rate, Body Weight, and BMI. This will be compared to FDA-cleared devices to determine equivalence: AtCor XCEL PWA & PWV to measure Pulse Wave Velocity and Pulse rate, and Detecto SOLO to measure Body Weight and BMI.
  Interventions: Device: PhysioWave Cardiovascular Analyzer; Device: AtCor XCEL PWA & PWV; Device: Detecto SOLO

INTERVENTIONS:
Device: PhysioWave Cardiovascular Analyzer — Measurement of Pulse Wave Velocity, Pulse Rate, Body Weight and BMI
Device: AtCor XCEL PWA & PWV — Measurement of Pulse Wave Velocity and Pulse Rate
Device: Detecto SOLO — Measurement of Body Weight and BMI

SUMMARY:
This is a prospective, single-center, non-randomized validation study being conducted under a non-significant risk study design with the primary aim to evaluate PWV, PR, and BW accuracy in a sample of subjects representative of the US general adult population. The primary study objective is to demonstrate equivalency when measuring: Pulse Wave Velocity (PWV) and Pulse Rate (PR) between the PhysioWave Cardiovascular Analyzer (CA) and AtCor Medical SphygmoCor® XCEL PWA & PWV (XCEL), and Body Weight (BW) between the CA and the Detecto Solo Digital Healthcare Scale (Detecto).

ELIGIBILITY:
Inclusion Criteria:

* Subjects >18 years old
* Subject signs a written Informed Consent form to participate in the study, prior to any study procedures

Subgroup Inclusion Criteria

* Subject has been taking ACE Inhibitors or Angiotensin Receptor Blockers for at least 30 days

Exclusion Criteria:

* Known significant carotid or femoral artery stenosis
* Non-palpable (non-detectable) arterial pulse at the sites of measurements
* Pacemaker, defibrillator, or other cardiac stimulator
* Erratic, accelerated or mechanically controlled irregular heart rhythm, or an arrhythmia
* History of cardiac valve disorder or cardiac valve disease
* History of venous disease, including venous insufficiency or deep vein thrombosis
* History of peripheral artery disease
* Requirement for supplemental oxygen
* Neuromuscular disorders that cause shaking or tremors (such as Parkinson's disease or Multiple Sclerosis), or other disease or condition affecting balance
* Amputation or malformation of any limb or extremity (foot, leg, or arm) which would impede the placement of blood pressure cuffs or standing on the scale with two feet.
* Known or suspected pregnancy
* Inability to provide informed consent
* Mental incompetence or a prisoner status
* Current participation in a clinical trial of another investigational drug or device in which the study endpoint has not been met
* BMI > 40
* Subjects > 400 lbs
* Subjects on strong vasoactive drugs, such as those used to control high blood pressure, for <30 days
* Blood loss or blood donation of ˃ 550 mL within 30 days before study procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2017-05-19 (Actual); Study Completion 2017-05-19 (Actual)

PRIMARY OUTCOMES:
Primary Objective: PWV Equivalence | Day 1
  The first primary study objective is to demonstrate equivalency when measuring: pulse wave velocity (PWV) (in m/s) between the PhysioWave Cardiovascular Analyzer and AtCor Medical SphygmoCor® XCEL PWA & PWV.
Pulse Rate Equivalence | Day 1
  The second primary study objective is to demonstrate equivalency when measuring: pulse rate (in bpm) between the PhysioWave Cardiovascular Analyzer and AtCor Medical SphygmoCor® XCEL PWA & PWV.
Body Weight Equivalence | Day 1
  The third primary study objective is to demonstrate equivalency when measuring body weight (in kg) between the PhysioWave Cardiovascular Analyzer and the Detecto Solo.

SECONDARY OUTCOMES:
Secondary Objective: BMI Equivalence | Day 1
  Demonstrate equivalency when measuring Body Mass Index (BMI) (in kg/m^2) between the PhysioWave Cardiovascular Analyzer and the Detecto Solo
Secondary Objective: Precision Analysis, PWV | Day 1 or Day 2
  Evaluate the precision of PWV measurements (in m/s) due to the sources of variation in measurements in the PhysioWave Cardiovascular Analyzer and AtCor Medical SphygmoCor® XCEL PWA & PWV. Sources of variation to be assessed include between-replicates, between-device, between-operator, and total (overall).
Secondary Objective: Precision Analysis, Pulse Rate | Day 1 or Day 2
  Evaluate the precision of pulse rate measurements (in bpm) due to the sources of variation in measurements in the PhysioWave Cardiovascular Analyzer and AtCor Medical SphygmoCor® XCEL PWA & PWV. Sources of variation to be assessed include between-replicates, between-device, between-operator, and total (overall).
Secondary Objective: Precision Analysis, Body Weight | Day 1 or Day 2
  Evaluate the precision of body weight measurements (in kg) due to the sources of variation in measurements in the PhysioWave Cardiovascular Analyzer and the Detecto Solo. Sources of variation to be assessed include between-replicates, between-device, between-operator, and total (overall).
Secondary Objective: Precision Analysis, BMI | Day 1 or Day 2
  Evaluate the precision of BMI measurements (in kg/m^2) due to the sources of variation in measurements in the PhysioWave Cardiovascular Analyzer and the Detecto Solo. Sources of variation to be assessed include between-replicates, between-device, between-operator, and total (overall).

OTHER OUTCOMES:
Exploratory Analysis: Impact of Strong Vasoactive Drugs on PWV Equivalence | Day 1
  An exploratory analysis will be conducted to evaluate any effects of strong vasoactive drugs, such as those used to control high blood pressure, on equivalency when measuring: pulse wave velocity (PWV) (in m/s) between the PhysioWave Cardiovascular Analyzer and AtCor Medical SphygmoCor® XCEL PWA & PWV.
Exploratory Analysis: Impact of BMI on PWV Equivalence | Day 1
  An exploratory analysis will be conducted to evaluate any effect(s) of BMI (in kg/m^2) on equivalency when measuring: pulse wave velocity (PWV) (in m/s) between the PhysioWave Cardiovascular Analyzer and AtCor Medical SphygmoCor® XCEL PWA & PWV.

CONTACTS AND LOCATIONS:
Locations (1):
- Diablo Clinical Research, Walnut Creek, California, United States

IPD SHARING:
Plan to Share IPD: No